CLINICAL TRIAL: NCT04615351
Title: A Pragmatic Approach to Lowering the Risk of Diabetes Mellitus After A Diagnosis of Gestational Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1248906-9
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Metformin 500 mg to be taken twice per day for two weeks and then metformin 1000 mg PO twice daily after tolerating the lower dose
  Interventions: Drug: Metformin
- Routine Care (No Intervention): Discharge information about maintaining a healthy diet

INTERVENTIONS:
Drug: Metformin — Medication
  Arms: Metformin

SUMMARY:
A Pilot of Metformin Postpartum

DETAILED DESCRIPTION:
The overall goal of this proposal is to assess metformin initiation at the time of hospital discharge for women with a history of gestational diabetes mellitus (GDM) improves maternal health at 1 year post-partum. Our central hypothesis is that diabetes mellitus (DM) prevention with metformin can be initiated days after delivery, rather than months to years after delivery, and result in a pragmatic and efficacious means of preventing DM and improving weight loss over the first year post-partum. To test this hypothesis, we will perform a open-label randomized controlled trial of metformin compared to placebo routine care initiated at the time of hospital discharge in women with a history of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Diabetes

Exclusion Criteria:

* Cannot tolerate metformin

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Prediabetes or Diabetes | 1 year postpartum
  glycosylated hemoglobin (HgbA1c) at 1 year postpartum (>/= 5.7% defined as prediabetes, >/=6.5% defined as DM

SECONDARY OUTCOMES:
Prediabetes or diabetes at 15 months postpartum | 15 months after delivery and study initiation
  HgbA1c at 15 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes